CLINICAL TRIAL: NCT07349225
Title: A Single-Arm, Multicenter, Prospective Phase II Clinical Study of Iparomlimab and Tuvonralimab Injection Combined With Chemotherapy and Sequential Thoracic Radiotherapy as First-Line Treatment for Extensive-Stage Small Cell Lung Cancer
Brief Title: Iparomlimab and Tuvonralimab Injection Combined With Chemotherapy and Sequential Thoracic Radiotherapy for Extensive-Stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-RE1-25001
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: ES-SCLC
MeSH Terms: interventions — Etoposide; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab Injection Combined with EP and Sequential Thoracic Radiotherapy (Experimental): Subjects first underwent induction therapy, receiving 4 to 6 cycles of Iparomlimab and Tuvonralimab Injection combined with etoposide and cisplatin. Upon completion of treatment, imaging evaluation was performed. Subjects who achieved a response of CR, PR, or SD with good local control proceeded to receive sequential thoracic radiotherapy (TRT), followed by maintenance therapy with Iparomlimab and Tuvonralimab Injection as a single agent.
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection; Drug: Etoposide; Drug: Cisplatin; Radiation: Targeted Radiation Therapy

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection — Induction Therapy: Ipilimumab and tuvonralimab injection, 5 mg/kg, Day 1, every 3 weeks for 4 to 6 cycles.
  Maintenance therapy: Ipilimumab and tuvonralimab injection, 5 mg/kg, Day 1, every 3 weeks. Maintenance therapy was continued for up to 2 years or until disease progression (PD), intolerable toxicity, withdrawal of informed consent, investigator-determined subject discontinuation from the study, non-compliance with study treatment or procedures, or other reasons specified in the protocol.
Drug: Etoposide — Induction Therapy: etoposide, 100 mg/m2, D1-3, every 3 weeks for 4 to 6 cycles.
Drug: Cisplatin — Induction Therapy: cisplatin, 25 mg/m², D1-3, every 3 weeks for 4 to 6 cycles.
Radiation: Targeted Radiation Therapy — Subjects who achieved a CR, PR, or SD with good local control following induction therapy, were subjected to sequential TRT (≥3Gy×10 or 15, using an involved-field irradiation technique. The specific regimen could be adjusted according to the patient's disease status and the standard practices of the investigator's institutional radiation oncology department)

SUMMARY:
This study will evaluate the efficacy and safety of Iparomlimab and Tuvonralimab Injection in combination with Chemotherapy and Sequential Thoracic Radiotherapy as First-Line Treatment for Extensive-Stage Small Cell Lung Cancer.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multicenter clinical study assessing the efficacy and safety of Iparomlimab and Tuvonralimab Injection in combination with Chemotherapy and Sequential Thoracic Radiotherapy as First-Line Treatment for Extensive-Stage Small Cell Lung Cancer. As well as, this study aimed to longitudinally monitor the dynamic changes of molecular residual disease in patients with extensive-stage small cell lung cancer to evaluate treatment efficacy and explore the potential application value of MRD as a biomarker for efficacy assessment.

ELIGIBILITY:
Inclusion Criteria:

1. For voluntary signing of the informed consent form, participants aged 18 to 75 years (inclusive), regardless of gender, are eligible
2. Histologically or cytologically confirmed ES-SCLC (according to the Veterans Administration Lung Study Group [VALG] staging system)
3. Expected survival ≥ 3 months
4. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
5. No prior systemic first-line therapy or immune checkpoint inhibitor treatment for ES-SCLC
6. Prior treatment with curative-intent surgery and adjuvant therapy (e.g., radiotherapy or chemotherapy), with a treatment-free interval of at least 6 months between the last dose of chemotherapy/radiotherapy/chemoradiotherapy and the diagnosis of ES-SCLC
7. According to RECIST v1.1 (Appendix 2), previously irradiated lesions can only be considered measurable if there is documented disease progression at that site after radiotherapy, and such lesions must not be the sole site of disease
8. Laboratory test results must meet the following criteria prior to enrollment: a) Hematology: No blood transfusion or hematopoietic growth factor administration within 14 days before enrollment; white blood cell count (WBC) ≥3.0×10^9/L; absolute neutrophil count (ANC) ≥1.5×10^9/L; platelets (PLT) ≥100×10^9/L; hemoglobin (HGB) ≥9.0 g/dL. b) Liver function: Non-liver metastasis subjects: Aspartate aminotransferase (AST) ≤2.5×ULN and alanine aminotransferase (ALT) ≤2.5×ULN. Liver metastasis subjects: ALT and AST ≤5×ULN; serum total bilirubin (TBIL) ≤1.5×ULN (except Gilbert syndrome, where TBIL ≤3.0 mg/dL). c) Renal function: Serum creatinine ≤1.5×ULN or calculated creatinine clearance (CrCl) ≥50 mL/min (using the Cockcroft-Gault formula in Appendix 3). d) Coagulation: International normalized ratio (INR) ≤1.5×ULN or activated partial thromboplastin time (APTT) ≤1.5×ULN (only for subjects not receiving anticoagulation therapy; subjects on stable-dose anticoagulants are eligible). e) Other tests confirming adequate cardiopulmonary function
9. Male patients with reproductive potential or female patients of childbearing potential must use effective contraception (e.g., oral contraceptives, intrauterine devices, or barrier methods combined with spermicides) during the study and continue for 6 months after treatment completion
10. For patients with HBV or HCV infection, the following criteria must be met: HBV-infected patients (HBsAg or HBV-DNA positive): Prior to the first treatment, HBV-infected patients must receive ≥3 days of guideline-recommended antiviral therapy with confirmed reduction in HBV-DNA levels upon retesting . Standard antiviral treatment must continue throughout the study period . HCV-infected subjects (HCVAb or HCV RNA positive): Must be in a stable condition as judged by the investigator. If already on antiviral therapy, treatment should be maintained during the study
11. Good compliance and cooperation with follow-up

Exclusion Criteria:

1. Patients with allergies or intolerance to the EP chemoradiotherapy regimen or any active/auxiliary components of the investigational drug
2. Active or untreated central nervous system (CNS) metastases identified by computed tomography (CT) or magnetic resonance imaging (MRI) during screening or prior radiographic assessments
3. Malignant effusions (pleural/ascites/pericardial) refractory to prior interventions (Defined as significant reaccumulation requiring repeat drainage or other interventions within 2 weeks, accompanied by symptomatic worsening)
4. Active autoimmune diseases , including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), inflammatory bowel disease (IBD), antiphospholipid syndrome, granulomatosis with polyangiitis (Wegener's), Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis (MS)
5. Uncontrolled hypertension despite treatment with ≥1 antihypertensive agent(s) (Defined as systolic blood pressure (SBP) ≥160 mmHg or diastolic blood pressure (DBP) ≥100 mmHg, based on the average of ≥2 BP readings, despite ongoing antihypertensive therapy. Adjustment of treatment to improve these parameters is permitted.)
6. Moderate-to-severe pulmonary diseases that significantly impair lung function , including but not limited to interstitial lung disease (ILD), drug-induced pneumonitis, idiopathic pneumonia, or idiopathic pulmonary fibrosis (IPF)
7. Patients with active tuberculosis infection confirmed by medical history or CT examination, or those with a history of active tuberculosis infection within 1 year prior to enrollment
8. Severe infections within 4 weeks prior to initial treatment , including but not limited to hospitalization due to infectious complications, bacteremia, or severe pneumonia
9. Severe cardiovascular or cerebrovascular diseases within 3 months prior to initial treatment , including myocardial infarction, cerebrovascular accident, unstable arrhythmia, or unstable angina
10. History of allogeneic bone marrow transplantation or solid organ transplantation
11. Prior treatment with immune checkpoint inhibitors (ICIs) , including but not limited to anti-PD-1, anti-PD-L1, or anti-CTLA-4 agents
12. Use of systemic immunosuppressive therapy within 2 weeks prior to initial treatment , or anticipated need for systemic immunosuppressive therapy during the study treatment period
13. Participation in any other interventional clinical study or use of any other investigational product within 4 weeks prior to signing the informed consent form
14. History of abdominal or tracheoesophageal fistula, gastrointestinal perforation, or intra-abdominal abscess within 1 month prior to initial treatment
15. Major vascular disease occurring within 3 months prior to initial treatment (e.g., aortic aneurysm requiring surgical repair)
16. Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study
17. Positive for human immunodeficiency virus (HIV) antibody
18. History of schizophrenia or psychotropic drug abuse
19. Other factors considered by the investigator to make the subject unsuitable for participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 1 year
  PFS was defined as the time from the first administration of the study drug to the first occurrence of objective tumor progression or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Objective Response Rate | 1 year
  ORR was defined as the proportion of patients whose best observed response from the first administration of the study drug until the first objective tumor progression was either CR (Complete Response) or PR (Partial Response).
Disease Control Rate | 1 year
  DCR was defined as the proportion of patients whose best observed response from the first administration of the study drug until the first objective tumor progression was CR, PR, or SD (Stable Disease).
Duration of Response | 1 year
  The time from the date of the first tumor assessment documenting CR or PR to the date of the first assessment documenting PD (Progressive Disease) or death from any cause, whichever occurred first, during the study treatment period.
Thoracic Local Control Rate | 1 year
  Defined as the proportion of patients who maintained control of the primary thoracic tumor and regional lymph nodes from the initiation of thoracic radiotherapy (TRT).
Overall Survival | 1 year
  The time from the first administration of the study drug to death from any cause.

IPD SHARING:
Plan to Share IPD: No